CLINICAL TRIAL: NCT02143115
Title: Comparative Effectiveness of Virtual and Optical Colonoscopy for Colorectal (CRC) Surveillance
Brief Title: Comparative Effectiveness of CTC & OC
Status: Completed | Type: Observational
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: R01CA155347 (NIH)
Record Dates: First submitted 2014-05-15; First posted 2014-05-20 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer surveillance
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Optical colonoscopy — Examination of the colon with a colonoscope
Radiation: CT-Colonography — A computerized X-ray that may find out if there are polyps or cancers and also pictures the contents of the abdomen and pelvis
  Other Names: CT-C or virtual colonoscopy

SUMMARY:
The goal of this study is to compare the findings of virtual (CT-colonography) with findings of optical colonoscopies to determine if virtual colonoscopy is suitable for colorectal cancer surveillance.

DETAILED DESCRIPTION:
The goal of this study is to compare, both clinically and from a cost-effectiveness perspective, virtual or CT-C (CT-Colonography) to standard CT scan and optical colonoscopy (OC). Virtual colonoscopy is a combination of a radiologic evaluation of the abdomen and pelvis with intra-colonic imaging. Previous research supports the concept that CT-C may be an effective substitute for the current OC and address limited compliance for surveillance for CRC survivors. Post-operative CRC surveillance strategies are effective, but depend upon patient compliance which is less than desired. Improved adherence is linked with greater cost-effectiveness as well as better clinical outcomes. CT-C possesses potential advantages: convenience as a single test, less risk, possibly patient preference and lower total costs. Costs would be reduced through direct (provision of fewer optical colonoscopies) and indirect means (reduction in time lost from work by patient and chaperone, etc.). When extrapolated across the roughly 200,000 OCs performed annually in the US for this indication reduced utilization of even 50% in a high unit cost procedure like OC would yield substantial savings without a reduction in clinical quality.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of CRC without clear evidence of metastatic disease who have completed their acute cancer-specific treatment
* Patients aged 18 years or older
* Patients who have signed an approved informed consent form

Exclusion Criteria:

* Patients with a diverting ileostomy, with a history of inflammatory bowel disease, FAP, or active GI symptoms (gastrointestinal bleed, diarrhea, severe abdominal pain, etc.)
* Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a history of colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2011-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Compare the test characteristics (sensitivity, specificity, positive and negative predictive value) of Computed Tomography colonography (CT-C) in the post Colorectal cancer resection using optical colonoscopy as the reference standard | One year post colorectal cancer resection
  To evaluate the test characteristics (sensitivity, specificity, positive and negative predictive value) of CT colonography (CT-C) for detecting colorectal adenomas and cancers in the post-CRC resection surveillance setting, using optical colonoscopy (OC) as the reference standard.

SECONDARY OUTCOMES:
Compare the costs and outcomes of Computed Tomography Colonography versus independent Optical Colonoscopy plus Computed Tomography for post Colorectal Cancer resection surveillance. | One year post colorectral cancer resection
  Compare the costs and outcomes, from third party payor and societal perspectives, of CT-C versus independent OC plus CT for post CRC resection surveillance, using standard methods of cost-effectiveness analysis.

CONTACTS AND LOCATIONS:
Overall Officials: David S Weinberg, MD, Principal Investigator — Fox Chase Cancer Center
Locations (5):
- United States (5):
  - University of Chicago, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weinberg DS, Mitnick J, Keenan E, Li T, Ross EA. Post-operative colorectal cancer surveillance: preference for optical colonoscopy over computerized tomographic colonography. Cancer Causes Control. 2019 Nov;30(11):1269-1273. doi: 10.1007/s10552-019-01231-w. Epub 2019 Sep 17. PMID 31531798
- [Derived] Kupfer SS, Lubner S, Coronel E, Pickhardt PJ, Tipping M, Graffy P, Keenan E, Ross E, Li T, Weinberg DS. Adherence to postresection colorectal cancer surveillance at National Cancer Institute-designated Comprehensive Cancer Centers. Cancer Med. 2018 Nov;7(11):5351-5358. doi: 10.1002/cam4.1678. Epub 2018 Oct 18. PMID 30338661
- [Derived] Weinberg DS, Pickhardt PJ, Bruining DH, Edwards K, Fletcher JG, Gollub MJ, Keenan EM, Kupfer SS, Li T, Lubner SJ, Markowitz AJ, Ross EA. Computed Tomography Colonography vs Colonoscopy for Colorectal Cancer Surveillance After Surgery. Gastroenterology. 2018 Mar;154(4):927-934.e4. doi: 10.1053/j.gastro.2017.11.025. Epub 2017 Nov 22. PMID 29174927